CLINICAL TRIAL: NCT04977427
Title: Dextenza vs Prednisolone Acetate After Cataract Surgery for Patients With Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Baylor Research Institute (Other)
Responsible Party: Principal Investigator, Jacob Fleenor, Resident Physician, Principal Investigator, Baylor Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iRIS RB Number 021-167
Record Dates: First submitted 2021-06-29; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Cataract Diabetic; Macula Edema
Keywords: Prednisolone; Dextenza
MeSH Terms: interventions — Calcium Dobesilate; prednisolone acetate

STUDY DESIGN:
Intervention Model Description: Randomized Fellow-Eye study design, in which one randomized eye in each patient undergoing bilateral cataract surgery receives standard prednisolone therapy, the other eye receiving the investigational Dextenza treatment.
Who Masked: Outcomes Assessor
Masking Description: Unable to fully mask to investigator in order to maintain safety (must assess the investigational Dextenza insert and its position in the lower punctum at each office visit).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prednisolone Arm (Active Comparator): Standard post-cataract surgery therapy arm; acts as control in each patient.
  Interventions: Drug: Prednisolone Acetate 1% Oph Susp
- Dextenza Arm (Active Comparator): Investigational arm to compare the effectiveness of the Dextenza insert to standard therapy.
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — Dexamethasone inserted into lower punctum at the end of cataract surgery in order to control inflammation in the eye for the following 30 days after surgery.
  Arms: Dextenza Arm
Drug: Prednisolone Acetate 1% Oph Susp — Standard Prednisolone taper following cataract surgery, QID for one week, followed by TID for one week, BID for one week, and QDaily for one week, then stop.
  Arms: Prednisolone Arm

SUMMARY:
This study aims to compare the effectiveness of Dextenza vs standard of care prednisolone taper after cataract surgery in diabetic patients with regards to controlling post-op inflammation at post-op days 7, 14, and 30.

DETAILED DESCRIPTION:
The inflammation after cataract surgery is controlled at the investigators' institution by a taper of prednisolone acetate 1%, which consists of four drops daily for one week, followed by three drops daily for one week, then two drops daily for one week, then one drop daily for one week. Due to the frequency of drops needed after cataract surgery, compliance with the post-op regimen often wavers. This study aims to evaluate the efficacy of Dextenza, which has been shown to be better than placebo after cataract surgery (1), against prednisolone acetate taper. If shown to be as effective without compromising safety, it could be a very convenient alternative to prednisolone acetate taper. Furthermore, if Dextenza is shown to be as effective as prednisolone taper in diabetic patients, it could be logically generalized that it would be effective in patients without diabetes as well, as patients without diabetes (and with no confounding risk factors, such as a history of uveitis) are less prone to developing post-op macular edema. Risks are minimal for this FDA approved treatment and include iridocyclitis (10%); intraocular pressure increased (6%); visual acuity reduced (2%); cystoid macular edema (1%); corneal edema (1%); eye pain (1%) and conjunctival hyperemia (1%). These risks are comparable to prednisolone acetate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed diabetes
* Patients must be undergoing cataract surgery in each eye
* Patients must have no worse than moderate nonproliferative diabetic retinopathy

Exclusion Criteria:

* Patients must not have any history of documented macular edema on OCT
* Patients must not have any macular edema on pre-op OCT
* Patients must not have any history of uveitis
* Patients must not have severe nonproliferative or proliferative diabetic retinopathy
* Patients with operative complications will be excluded from this study
* Patients with any active corneal disease, infectious or rheumatologic, will be excluded
* Patients must not be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Intraocular Inflammation | 7 days
  The investigators will assess the effect of 0.4mg dexamethasone intracanalicular insert on the presence or absence of inflammation in the eye following cataract surgery when compared to prednisolone acetate 1%.
Intraocular Inflammation | 14 days
  The investigators will assess the effect of 0.4mg dexamethasone intracanalicular insert on the presence or absence of inflammation in the eye following cataract surgery when compared to prednisolone acetate 1%.
Intraocular Inflammation | 30 days
  The investigators will assess the effect of 0.4mg dexamethasone intracanalicular insert on the presence or absence of inflammation in the eye following cataract surgery when compared to prednisolone acetate 1%.

SECONDARY OUTCOMES:
Macular Edema | 7 days
  The investigators will assess the effect of 0.4mg dexamethasone intracanalicular insert on the presence or absence of macular edema in the eye on OCT imaging following cataract surgery when compared to prednisolone acetate 1%.
Macular Edema | 14 days
  The investigators will assess the effect of 0.4mg dexamethasone intracanalicular insert on the presence or absence of macular edema in the eye on OCT imaging following cataract surgery when compared to prednisolone acetate 1%.
Macular Edema | 30 days
  The investigators will assess the effect of 0.4mg dexamethasone intracanalicular insert on the presence or absence of macular edema in the eye on OCT imaging following cataract surgery when compared to prednisolone acetate 1%.

IPD SHARING:
Plan to Share IPD: No